CLINICAL TRIAL: NCT00171301
Title: 1-year Extension to CICL670A2402 an Open-label, Multi-center Trial of the Efficacy and Safety of Long-term Treatment With Deferasirox (10 to 20 mg/kg/Day) in Beta-thalassemia Patients With Transfusional Hemosiderosis (Study Amended to 2- Year Duration)
Brief Title: Extension Study of the Efficacy and Safety of Deferasirox Treatment in Beta-thalassemia Patients With Transfusional Hemosiderosis (Study Amended to 2-year Duration)
Acronym: ESCALATOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2402E1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Beta-thalassemia Major; Hemosiderosis; Iron Overload; Rare Anemia
Keywords: Transfusional hemosiderosis; Beta-thalassemia major; Deferasirox; iron overload; rare anemia; iron overload due to transfusion
MeSH Terms: conditions — beta-Thalassemia; Hemosiderosis; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deferasirox (Experimental): Deferasirox was given orally once daily (10 to 20 mg/kg) to participants 2 years and older based on participant's body weight.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferasirox was administered orally once daily. Deferasirox was available as 125 mg, 250 mg, and 500 mg tablets.
  Other Names: Exjade

SUMMARY:
To allow patients treated with deferasirox in the core study to continue iron chelation therapy for 2 years or until the drug became locally commercially available. To evaluate the long-term safety and efficacy of deferasirox by measuring treatment success, change in liver iron content (LIC) and change in serum ferritin levels. Safety was mainly assessed by incidence of adverse events (AEs)and clinically significant lab parameters.

DETAILED DESCRIPTION:
Iron accumulation is an inevitable consequence of chronic blood transfusions and results in serious complications in the absence of chelation treatment to remove excess iron. Deferasirox (Exjade, ICL670) is an oral chelator with high iron-binding potency and selectivity. This extension study aimed at collecting efficacy and safety data during 2 years of treatment with deferasirox in the extension study or until deferasirox became commercially available in the countries where the centers were located, whichever came first. The population comprised of β-thalassemia patients with transfusional hemosiderosis who could not be satisfactorily treated with deferoxamine or deferiprone.

ELIGIBILITY:
Inclusion Criteria:

* Patients completing the planned 12-month core study (NCT00171171)
* Female patients who have reached menarche and who are sexually active must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation
* Written informed consent obtained from the patient and/or legal guardian on the patient's behalf in accordance with the national legislation

Exclusion Criteria:

* Pregnant or breast feeding patients.
* Patients being considered by the investigator potentially unreliable and/or not cooperative with regard to the core study protocol, or the planned extension protocol

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Cairo, Egypt
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Muscat, Oman
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Damascus, Syria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an Extension to Core Study CICL670A2402 (NCT00171171). 233 participants completed the core study and entered this extension study.
Pre-assignment Details: 2 participants from the 16 and older group did not receive deferasirox. Thus, the 16 and older group comprises of 69 treated participants.
Groups:
- Deferasirox (Between 2 <16 Years ): Participants age 2 years up to 16 years received a daily oral dose of deferasirox. Dose selection was based on the dose last received in the core study. The individual daily doses of deferasirox and the exact amount of tablets (125, 250, or 500 mg) contributing to each dose were calculated by the investigator based on the patient's body weight.
- Deferasirox (16 Years or Older): Participants age 16 years or older received a daily oral dose of deferasirox. Dose selection was based on the dose last received in the core study. The individual daily doses of deferasirox and the exact amount of tablets (125, 250, or 500 mg) contributing to each dose were calculated by the investigator based on the patient's body weight.
Period: Overall Study
Arm/Group | Deferasirox (Between 2 <16 Years ) | Deferasirox (16 Years or Older)
Started | 162 | 71 (2 participants in this group never received deferasirox.)
Received Deferasirox | 162 | 69
Completed | 154 | 62
Not Completed | 8 | 9
Not completed — Death | 1 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 6 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox (Between 2 <16 Years ) | Deferasirox (16 Years or Older) | Total
Number analyzed (Participants) | 162 | 71 | 233
Age Continuous [Mean (Standard Deviation); unit: years] — Safety Population consisting of all participants who received study drug in the Extension study n= 231.
  years | 9.5 (3.59) | 21.2 (5.82) | 13.0 (6.93)
Sex/Gender, Customized [Number; unit: participants] — Safety Population consisting of all participants who received study drug in the Extension study n=231.
  participants
    Female | 80 | 35 | 115
    Male | 82 | 36 | 118

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success From Core Baseline (BL) to Extension End of Study, by Baseline LIC Level and Age
Description: Success was defined as the percentage of participants with decreased liver iron content (LIC) at the end of extension study compared to core baseline (BL) LIC. Success Criteria: For participants with Baseline LIC from 1 - <7 mg Fe/g dw, success was achieved if LIC level maintained at 1 - <7 mg Fe/g dw. For participants with Baseline LIC ≥7 - <10 mg Fe/g dw, success was achieved if LIC dropped to between 1 and < 7 mg Fe/g dw. For participants with Baseline LIC ≥10 mg Fe/g dw, success was achieved if LIC dropped by at least 3 mg Fe/g dw. LIC was measured by biopsy or magnetic resonance imaging.
Time Frame: From Core Study Baseline, to Extension End of Study, Up to 3 Years
Population: The primary analysis will be on the intent-to-treat (ITT) population. ITT population includes all participants who performed the core end of study (EOS) visit evaluation and assessments and were included in the extension study. "n" is the number of participants analyzed in each category.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Deferasirox (Between 2 <16 Years): Participants age 2 years up to 16 years received a daily oral dose of deferasirox. Dose selection was based on the dose last received in the core study. The individual daily doses of deferasirox and the exact amount of tablets (125, 250, or 500 mg) contributing to each dose were calculated by the investigator based on the patient's body weight.
Arm/Group | Deferasirox (Between 2 <16 Years) | Deferasirox (16 Years or Older)
Number analyzed (Participants) | 162 | 71
percentage of participants
  Core Baseline LIC 1-<7 mg Fe/g dw (n=20, 2) | 75.0 [56.0 to 94.0] | 100 [15.8 to 100]
  Core Baseline LIC 7-<10 mg Fe/g dw (n=18, 8) | 72.2 [51.5 to 92.9] | 50.0 [15.7 to 84.3]
  Core Baseline LIC ≥10 mg Fe/g dw (n=124, 61) | 76.6 [69.2 to 84.1] | 73.8 [62.7 to 84.8]

2. Primary Outcome: Absolute Change in Liver Iron Concentration (LIC)Measured by Liver MRI or Liver Biopsy From Core Study Baseline (BL) to End of Extension Study, by LIC Category
Description: Liver MRI or Liver Biopsy was performed at the core study baseline (BL) and then 1 year and 2 years in the core study, baseline of the extension study and time of discontinuation from the extension visit (end of study). Liver iron content (LIC) is reported in milligram Iron per gram dry weight (mg Fe/g dw).
  Absolute change in LIC from core study baseline to the end of the extension study is presented for participants with the following two core study baseline LIC levels: 1-<7 mg Fe/g dw and ≥7 mg Fe/g dw.
Time Frame: From Baseline of Core Study to End of Extension Study, up to 3 years
Population: Participants from the Intent-to-Treat (ITT) population for whom LIC data was available at Core Study baseline and at the End of Extension Study. "n" is the number of participants analyzed in each category.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox (Between 2 <16 Years) | Deferasirox (16 Years or Older)
Number analyzed (Participants) | 119 | 41
mg Fe/g dw
  Core Baseline LIC 1-<7 mg Fe/g dw (n=12, 0) | -1.32 (3.125) | NA (NA) — No participants in this category for this group.
  Core Baseline LIC ≥7 mg Fe/g dw (n=107, 41) | -9.03 (9.260) | -8.39 (11.312)

3. Secondary Outcome: Absolute Change in Serum Ferritin Level Measured From Core Study Baseline (BL) to End of Extension Study
Description: Serum Levels were assessed at core study baseline (BL), 1 year, 2 years in core study, baseline of extension study and time of discontinuation from the extension visit (end of study) in monthly intervals. Serum Ferritin is reported in micrograms per Liter (µg/L).
Time Frame: From Baseline of Core Study to End of Extension Study, up to 3 years
Population: Participants from the Intent-to-Treat (ITT) population for whom Serum Ferritin data was available at Core Study baseline and at the End of Extension Study.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Deferasirox (Between 2 <16 Years) | Deferasirox (16 Years or Older)
Number analyzed (Participants) | 120 | 43
µg/L | -1432.51 (1969.622) | -1791.91 (2712.334)

4. Secondary Outcome: Absolute Change in Serum Ferritin Level for All Participants Measured From Core Study Baseline (BL) to End of Extension Study, by Baseline Liver Iron Content (LIC)
Description: Serum Levels were assessed at core study baseline (BL) and then 1 year and 2 years in core study, baseline of extension study and time of discontinuation from the extension visit (end of study). Serum Ferritin is reported in micrograms per Liter. Absolute change in Serum Ferritin from core study baseline to the end of the extension study is presented for participants with the following two core study baseline LIC levels: 1-<7 mg Fe/g dw and ≥7 mg Fe/g dw.
Time Frame: From Baseline of Core Study to End of Extension Study, up to 3 years
Population: Participants from the Intent-to-Treat (ITT) population for whom Serum Ferritin data was available at Core Study baseline and at the End of Extension Study. "n" is the number of participants analyzed in each category.
Measure: Mean (Standard Deviation); unit: µg/L
Groups:
- Deferasirox (All Participants): Participants received a daily oral dose of deferasirox. Dose selection was based on the dose last received in the core study. The individual daily doses of deferasirox and the exact amount of tablets (125, 250, or 500 mg) contributing to each dose were calculated by the investigator based on the patient's body weight.
Arm/Group | Deferasirox (All Participants)
Number analyzed (Participants) | 163
µg/L
  Core Baseline LIC 1-<7 mg Fe/g dw (n=12) | -369.83 (1349.57)
  Core Baseline LIC ≥ 7 mg Fe/g dw (n=151) | -1619.31 (2217.104)

ADVERSE EVENTS:
Time Frame: From baseline to end of study, up to 2 years
Description: Adverse Events were calculated for the Safety Population consisting of all participants who received study drug in this Extension study. (162 participants between 2 < 16 years, 69 participants 16 years or older. Total 231 participants in Safety Population.)
Groups:
- Deferasirox (16 Years or Older): Participants age 16 years and older received a daily oral dose of deferasirox. Dose selection was based on the dose last received in the core study. The individual daily doses of deferasirox and the exact amount of tablets (125, 250, or 500 mg) contributing to each dose were calculated by the investigator based on the patient's body weight.
Arm/Group | Deferasirox (Between 2 <16 Years) | Deferasirox (16 Years or Older)
Serious Adverse Events (participants affected / at risk) | 5/162 | 12/69
Other Adverse Events (participants affected / at risk) | 54/162 | 33/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (Between 2 <16 Years) (N=162) | Deferasirox (16 Years or Older) (N=69)
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Perinephric abscess (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 3
Blood creatinine increased (Investigations) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (Between 2 <16 Years) (N=162) | Deferasirox (16 Years or Older) (N=69)
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 17 | 5
Pain (General disorders) | 0 | 5
Pyrexia (General disorders) | 3 | 6
Gastroenteritis (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 26 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 8
Alanine aminotransferase increased (Investigations) | 13 | 4
Blood calcium decreased (Investigations) | 0 | 4
Blood creatinine increased (Investigations) | 5 | 9
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
An internal review revealed major Good Clinical Practice violations at 2 sites in Saudi Arabia: 602 for core + extension, 601 for 2-yr extension. Therefore data was excluded (completely for 602 + partly for 601) from analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.